CLINICAL TRIAL: NCT01117532
Title: Brief Group Intervention Using EFT (Emotional Freedom Techniques) for Depression in College Students: A Randomized Controlled Trial
Brief Title: Brief Group Intervention Using EFT (Emotional Freedom Techniques) for Depression in College Students
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Dawson Church, Executive Director, Soul Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMI-DEP-5410
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Depression
Keywords: students,; depression,; group therapy,; EFT (Emotional Freedom Techniques),; energy psychology
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EFT (Experimental): Four 90 minute group EFT classes
  Interventions: Behavioral: EFT (Emotional Freedom Techniques)
- No Treatment (No Intervention)

INTERVENTIONS:
Behavioral: EFT (Emotional Freedom Techniques) — Four 90 minute group therapy classes of this behavioral intervention
  Arms: EFT

SUMMARY:
Depression is an important mental health concern in college students. This study will recruit students who test positive for moderate to severe depression on the Beck Depression Inventory (BDI). Subjects will be randomly assigned to either a treatment or a control condition. Those in the treatment group will receive four 90 minute group classes using EFT (Emotional Freedom Techniques) to address traumatic memories and other self-identified causes of depression. It will compare them to a no treatment control group.

ELIGIBILITY:
Inclusion Criteria:

* A score of 19 or more on the Beck Depression Inventory
* Currently enrolled at the University of Santo Tomas
* Able to read, understand, and complete forms

Exclusion Criteria:

* None

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Student scores on the Beck Depression Inventory (BDI) | One month

CONTACTS AND LOCATIONS:
Locations (1):
- College of Science, University of Santo Tomas, Manila, Philippines

REFERENCES:
- [Result] Church D, De Asis MA, Brooks AJ. Brief group intervention using emotional freedom techniques for depression in college students: a randomized controlled trial. Depress Res Treat. 2012;2012:257172. doi: 10.1155/2012/257172. Epub 2012 Jul 17. PMID 22848802
- See also: National Institute for Integrative Healthcare — http://www.NIIH.org